CLINICAL TRIAL: NCT04596007
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HEC83518 Tablets in Chinses Healthy Subjects
Brief Title: The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of HEC83518 Tablets in Chinses Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC83518-P-01 / CRC-C1934
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All are double-blind except the pre-trial group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEC83518 tablets (Experimental): There will be a total of 7 dose cohorts: 5 mg,10 mg, 20 mg, 40 mg, 80 mg, and 140 mg,200 mg.
  Interventions: Drug: HEC83518 tablets
- placebo tablets (Placebo Comparator): There will be a total of 6 dose cohorts: 10 mg, 20 mg, 40 mg, 80 mg, and 140 mg,200 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC83518 tablets — Each dose of HEC83518 and placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  Arms: HEC83518 tablets
Drug: Placebo — placebo
  Arms: placebo tablets

SUMMARY:
The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of HEC83518 Tablets in Chinses Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
2. Without Plann for pregnancy or pregnant within 3 months after enrollment throughout the trial.
3. Subjects aged between 18 and 45 (both inclusive) years old.
4. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18 and ≤28 kg/m2 at screening.
5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
2. Subjects with history of digestive system,urinary system, liver,central nervous system, blood system, endocrine system,respiratory system,immune system,cardiovascular system,and/or malignant tumor or others medical conditions (such as history of mental illness, etc.) that are not suitable for clinical trial participation;Subjects with history of stroke, epilepsy, bipolar disorder/mania, high intraocular pressure, or acute angular-closure glaucoma.
3. Subjects with history of sleep-related illness.
4. Subjects with history of severe involuntary hypoglycemia
5. Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s) ,or anaphylaxis physique.
6. Use of any prescription or non-prescription medications within 14 days prior to initial dosing,or Use of any medications known to inhibit or induce cytochrome P enzyme drug metabolism within 28 days prior to initial dosing.
7. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
8. Positive results from urine drug screen test.
9. History of alcoholism or drink regularly within 3 months prior to the study(defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test.
10. Regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug.
11. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
12. Subjects who plan to receive or have had organ transplants.
13. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential.
14. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
15. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
The Number of Adverse Events (AEs) | up to 5 days
  Safety and Tolerability of HEC83518 by Assessment of the Number of Adverse Events (AEs) Following Administration in Single Ascending Dose .

SECONDARY OUTCOMES:
PK parameters - AUC0-∞ | up to 96 hours
  area under the concentration versus time curve (AUC) from time zero to infinity
PK parameters - Cmax | up to 96 hours
  Geometric Mean of Maximum Observed Plasma Concentration of HEC83518
PK parameters -tmax | up to 96 hours
  time to peak
PK parameters -t½ | up to 96 hours
  apparent terminal elimination half-life
PK parameters -Vz/F | up to 96 hours
  apparent volume of distribution
PK parameters - MRT | up to 96 hours
  the Mean Residence Time
PK parameters -CL/F | up to 96 hours
  the Apparent Clearance

OTHER OUTCOMES:
The pharmacodynamics of HEC83518 tablets | up to 24 hours
  The pharmacodynamics of HEC83518 was preliminarily explored through KSS (Karolinska sleepiness Scale, Karolinska Sleepiness Scale) and sleep monitoring instrument

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai xuhui district central hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No